CLINICAL TRIAL: NCT03403010
Title: A Randomized Cross-over Design Evaluating the Effects of Using a Rehabilitation-specific Gaming Software Platform for the Achievement of Individual Physiotherapy Goals of Children With Severe Spastic Cerebral Palsy.
Brief Title: Rehabilitation Specific Gaming in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vrije Universiteit Brussel (Other); Fondation Motrice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: s59104
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Children are randomized into the intervention group (conventional, usual therapy including the use of rehabilitation-specific gaming) or the control group (PT, usual physiotherapy not including gaming), followed by a cross-over. After the intervention period of 3 months, wash-out period will be organized to evaluate follow-up effects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control period (No Intervention): In this group conventional physiotherapy of the child will be continued and the therapist will be asked not to use any gaming activities. Also during the control period, the frequency and duration of the therapy sessions will not be influenced by the researchers.
- Intervention period (Active Comparator): In this group the usual individual physiotherapy program of the child will be continued as performed before the study and will be executed by the child's usual, familiar physiotherapist. The therapist will be asked to use the rehabilitation-specific gaming software every therapy session, for at least 15 to 20 minutes. The therapist will receive an extensive introduction and demonstration of the software and the researchers will participate in at least one therapy session.
  Interventions: Other: Rehabilitation-specific gaming platform
- Wash-out period (No Intervention): The wash-out period is considered after each intervention period. As during the control period, therapy will be continued as usual during the washout-period but no gaming is allowed during therapy.

INTERVENTIONS:
Other: Rehabilitation-specific gaming platform — The rehabilitation specific gaming software was developed as part of the ICT4rehab project with partners from the Vrije Universiteit Brussel and the University Libre de Bruxelles. The ICT4Rehab puts several ICT tools supporting 2/3D user interaction into place. The games can be controlled using a Kinect camera system (Microsoft(®) (Redmond, WA) Kinect™) or a Wii balance board (® NintendoTM, Japan), depending on the choice of the therapist and the needs of the child.
  Arms: Intervention period

SUMMARY:
The aim of this project is to evaluate the effectiveness of using rehabilitation-specific gaming in physical therapy of children with cerebral palsy.

The primary goal of this project is to evaluate the effectiveness of integrating 15 to 20 minutes of gaming using a rehabilitation-specific gaming platform into standard physiotherapy sessions on the achievement of individual goals of children with bilateral spastic cerebral palsy with GMFCS level III-IV.

The secondary goal of this project is to evaluate the effectiveness of integrating 15 to 20 minutes of gaming using a rehabilitation-specific gaming platform into standard physiotherapy sessions on trunk control and gross motor function of children with bilateral spastic cerebral palsy with GMFCS level III-IV.

DETAILED DESCRIPTION:
Forty children are recruited via the Cerebral Palsy Reference Centre (University Hospital Leuven, Pellenberg). Children are recruited when they have been diagnosed with bilateral spastic CP, Gross Motor Function Classification (GMFCS) level III-IV, aged between 6 and 15y and standardly receive physiotherapy at an intensity of minimally 2 times per week, 45 minutes per session.

Children are randomized into the intervention group (conventional, usual therapy including the use of rehabilitation-specific gaming) or the control group (PT, usual physiotherapy not including gaming), followed by a cross-over. After the intervention period of 3 months, wash-out period will be organized to evaluate follow-up effects.

During the intervention period, the usual individual physiotherapy program of the child will be continued as performed before the study and will be executed by the child's usual, familiar physiotherapist. The therapist will be asked to use the rehabilitation-specific gaming software every therapy session, for at least 15 to 20 minutes. The therapist will receive an extensive introduction and demonstration of the software and the researchers will participate in at least one therapy session.

During the control period, the usual, conventional physiotherapy of the child will be continued and the therapist will be asked not to use any gaming activities. Also during the control period, the frequency and duration of the therapy sessions will not be influenced by the researchers.

A wash-out period in between both programs, assumes that therapy effects are still present for a certain period after the intervention and therefore aims to wash-out these effects. Therefore, this period is considered after each intervention period. As during the control period, therapy will be continued as usual during the washout-period but no gaming is allowed during therapy.

All intervention and control periods will have the same duration of 3 months. During all periods, therapists will receive a diary to register the exact amount of therapy performed. The diary that will be provided during the intervention, will also question the specific games played and will register the therapy goals strived for.

Children will be evaluated before and after each intervention or control period using a multidimensional assessment protocol. In addition, children will also receive a follow-up evaluation 3 months after the last intervention period. This will result in 4 evaluation moments for each child. The evaluation exist of the Goal Attainment Scale, the Gross Motor Function Measure, the Pediatric Balance Scale, the Trunk Control Measurement Scale and the Dimensions of Mastery Motivation Questionnaire (DMQ).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Spastic CP
* Gross Motor Function Classification (GMFCS) level III-IV,
* Aged between 6 and 15y
* Standardly receive physiotherapy at an intensity of minimally 2 times per week, 45 minutes per session.

Exclusion Criteria:

* received multilevel surgery in the previous year
* IQ <70
* visual acuity <3/10

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scale (GAS) | 3 months
  Evaluates the achievement of the individual goals per child and allows comparison of a heterogeneous group of children. GAS is essentially conducted on a 5-point measure, with the degree of attainment captured for each goal area. If the patient achieves the expected level, this is scored at 0. If they achieve a better than expected outcome this is scored at: +1 (Somewhat better), +2 (much better). If they achieve a worse than expected outcome this is scored at: -1 (Somewhat worse) or -2 (much worse). Goals may be weighted to take account of the relative importance of the goal to the individual, and/or the anticipated difficulty of achieving it. Overall Goal Attainment Scores are then calculated by applying a formula. The composite GAS (the sum of the attainment levels x the relative weights for each goal) is transformed into a standardised measure or T score with a mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | 3 months
  The static subsection of the TCMS evaluates static trunk control during movements of upper and lower limbs. The dynamic section the TCMS evaluates the ability to perform active trunk movements in different planes within and beyond the base of support. The total scale contains 15 items, with the subscale consisting of 5, 7 and 3 items, respectively. All items are scored on a two-, three- or four-point ordinal scale and administered bilaterally in case of clinical relevance. The total score of the TCMS ranges from 0 to 58, with a higher score indicating a better performance.
Pediatric Balance Scale (PBS) | 3 months
  The PBS is a modification of the Berg Balance Scale, developed as a measure for children. It measures balance functions for school-aged children and provides clinicians with a standardized format for measuring performance of functional balance tasks ranging from timed sitting balance to standing on one leg. There is a total of 14 items, each item is scored utilizing the 0 to 4 scale. The child's performance should be scored based upon the lowest criteria, which describes the child's best performance. If on the first trail a child receives the maximal socre of 4, additional trails need not to be administered.
Gross Motor Function Measure-88 (GMFM) | 3 months
  The GMFM is a standardized observation measure to evaluate gross motor function changes in children with CP. It is divided into five difference dimensions, ranging from lying and rolling to jumping and running. There is a total of 88 items, each item is scored using a 4-point Likert scale. Values of 0 to 3 are assigned to the four categories: 0= does not initiate, 1=initiates, 2=partially completes and 3=completes. Each of the dimensions of the GMFM has a different number of items. Each dimension contributes equally to the total score, therefore a percent score can be calculated for each dimension. A total score is obtained by calculating the mean of five dimension scores.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No